CLINICAL TRIAL: NCT06155526
Title: Muscle Mechanical Response in Active vs. Passive Resting Exercise
Brief Title: Muscle Mechanical Response in Exercise.
Status: Completed | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Other Study IDs: 24112023
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Muscle Weakness
Keywords: tensiomyography; triceps; dorsal; exercise; pectoral
MeSH Terms: conditions — Muscle Weakness; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- active rest: patients taking an active rest after swimming sets
  Interventions: Other: Activity
- passive rest: patients taking a passive rest after swimming sets

INTERVENTIONS:
Other: Activity — patients taking an active rest after swimming sets
  Groups: active rest

SUMMARY:
The muscular response on the main muscles of the propulsive phase of the upper limb in crawl has been evaluated by tensiomyography (TMG), which was carried out through three parameters: activation time (Td), contraction time (Tc) and maximum deformation (Dm).

The objective of this study is to evaluate the hypothesis of changes produced between lactic resistance training with passive rest and lactic resistance training with active rest.

For this, thirty swimmers participated, with an average age of 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 25 years old.
* have a minimum mark or have participated by ranking in a crawl event in the territorial championship of Madrid in the current season belong.
* to the male gender.

Exclusion Criteria:

* subjects who did not meet the minimum age and did not obtain the minimum mark and did not sign the informed consent.

Ages: 18 Years to 25 Years | Sex: Male
Age Groups: Adult
Study Population: male swimmers from 18 to 25 years old with a minimum mark who swimming a croll style
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
activation time | 15 minutes
  activation time measured by tensomiography
contraction time | 15 minutes
  contraction time measured with tensomiography
maximum deformation | 15 minutes
  maximum deformation measured with tensomiography

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge V Velázquez Saornil, Ávila, Avila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palma, S., Silva, H., Gamboa, H., & Mil-Homens, P. (2008). Standing Jump Loft Time Measurement - An Acceleration based Method. International Conference on Bio-inspired Systems and Signal Processing.
- [Background] Cular D, Babic M, Zubac D, Kezic A, Macan I, Peyre-Tartaruga LA, Ceccarini F, Padulo J. Tensiomyography: from muscle assessment to talent identification tool. Front Physiol. 2023 Jun 26;14:1163078. doi: 10.3389/fphys.2023.1163078. eCollection 2023. PMID 37435303
- [Background] Gil S, Loturco I, Tricoli V, Ugrinowitsch C, Kobal R, Abad CC, Roschel H. Tensiomyography parameters and jumping and sprinting performance in Brazilian elite soccer players. Sports Biomech. 2015 Sep;14(3):340-50. doi: 10.1080/14763141.2015.1062128. Epub 2015 Aug 14. PMID 26271313
- [Background] Maloney SJ, Fletcher IM. Lower limb stiffness testing in athletic performance: a critical review. Sports Biomech. 2021 Feb;20(1):109-130. doi: 10.1080/14763141.2018.1460395. Epub 2018 May 16. PMID 29768094
- [Background] Douglas J, Pearson S, Ross A, McGuigan M. Reactive and eccentric strength contribute to stiffness regulation during maximum velocity sprinting in team sport athletes and highly trained sprinters. J Sports Sci. 2020 Jan;38(1):29-37. doi: 10.1080/02640414.2019.1678363. Epub 2019 Oct 19. PMID 31631783